CLINICAL TRIAL: NCT02186977
Title: Proof Of Concept Study: Immunogenicity and Safety of Hepatitis B Injection in the Dermis in Healthy Volunteers Using an Intradermal Injection Device (VAX-ID)
Brief Title: Proof Of Concept : Immunogenicity and Safety of hepB Injection in the Dermis Using VAX-ID
Acronym: POC_VAX-ID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novosanis NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CP140465_2014_001_v5
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B
Keywords: immunogenicity; safety; proof of concept
MeSH Terms: conditions — Hepatitis B | interventions — Injections, Intradermal; Injections, Intramuscular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intramuscular group (Active Comparator): These subjects will receive one intramuscular injection of 1.0cc HBVAXPRO 10mcgr/ml (Sanofi Pasteur-MSD) with syringe and needle in the deltoid region.
  Interventions: Drug: 1.0 cc HBVAXPRO 10mcgr/ml (Sanofi Pasteur MSD)
- Intradermal group (Mantoux) (Experimental): These subjects will receive one intradermal injection with mantoux technique in the forearm. 0.1cc of HBVAXPRO 40mcgr/ml (Sanofi Pasteur-MSD) will be injected.
  Interventions: Drug: 0.1cc HBVAXPRO 40mcgr/ml (Sanofi Pasteur MSD)
- Intradermal group (VAX-ID) A (Experimental): These subjects will receive one intradermal injection with the newly developed intradermal injection device VAX-ID in the forearm. 0.1cc of HBVAXPRO 40mcgr/ml (Sanofi Pasteur MSD) will be injected.
  Interventions: Device: VAX-ID
- Intradermal group (VAX-ID) B (Experimental): These subjects will receive two intradermal injections with two newly developed intradermal injection devices VAX-ID in both forearms each 0.1cc of HBVAXPRO 40mcgr/ml (Sanofi Pasteur MSD) will be injected.
  Interventions: Device: VAX-ID

INTERVENTIONS:
Device: VAX-ID — 0.1cc HBVAXPRO 40mcgr/ml (Sanofi Pasteur MSD) with each injection
  Other Names: INTRADERMAL
  Arms: Intradermal group (VAX-ID) A; Intradermal group (VAX-ID) B
Drug: 1.0 cc HBVAXPRO 10mcgr/ml (Sanofi Pasteur MSD) — 1.0 cc HBVAXPRO 10mcgr/ml (Sanofi Pasteur MSD)
  Other Names: INTRAMUSCULAR
  Arms: Intramuscular group
Drug: 0.1cc HBVAXPRO 40mcgr/ml (Sanofi Pasteur MSD) — 0.1cc HBVAXPRO 40mcgr/ml (Sanofi Pasteur MSD) with each injection
  Other Names: MANTOUX_INTRADERMAL
  Arms: Intradermal group (Mantoux)

SUMMARY:
A proof of concept (POC) study will be conducted in 44 volunteers that have been fully vaccinated against hepatitis B in the past (at least 5 years ago) to assess the safety and immunogenicity of intradermal vaccination with hepatitis B surface vaccine antigen using a newly developed intradermal injection device VAX-ID, compared to intramuscular and intradermal (Mantoux technique) injection.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults, checked anamnestically (based on medical history) at entry of the study
* 18-35 years
* vaccination status: fully vaccinated against hepatitis B at least 5 years ago, with proof of vaccine response (to avoid non-response among the subjects). Subjects has to ask for a document of this proof at the service occupational medicine of the University of Antwerp.
* capable of understanding, reading and writing Dutch

Exclusion Criteria:

* other vaccination(s) 4 weeks before study onset
* pregnancy and lactation (women will be questioned during anamnesis)
* plan to have other vaccination during the study period

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Anamnestic response after intradermal or intramuscular hepatitis B booster vaccination in previously fully immunized subjects | after 14 days

SECONDARY OUTCOMES:
Safety: solicited local and systemic reactions, unsolicited adverse events and Serious Adverse Events occurrence, intensity and relationship to vaccination of all Adverse Events reported during the 14-day follow-up period after the challenge dose | during 14 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, Prof, Principal Investigator — Centre for the Evaluation of Vaccination Vaccine & Infectious Disease Institute
Locations (1):
- Centre for the Evaluation of Vaccination Vaccine & Infectious Disease Institute, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No